CLINICAL TRIAL: NCT03729297
Title: The Efficacy of Cabozantinib in Advanced SAlivary Gland Cancer Patients, a Phase II Clinical Trial
Brief Title: Cabozantinib in Advanced Salivary Gland Cancer Patients
Acronym: Cabo ASAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: safety issues
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOHN14
Record Dates: First submitted 2018-07-24; First posted 2018-11-02 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2019-11

CONDITIONS: Salivary Gland Cancer
Keywords: salivary gland cancer; adenoid cystic carcinoma; salivary duct carcinoma; cabozantinib; progression free survival; overall survival; phase 2 clinical trial
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: 3 cohorts:
  * adenoid cystic carcinoma
  * salivary duct carcinoma
  * other subtypes of salivary gland cancer
  sample size: The Simon two-stage design will be used, The first stage consists of 9 patients per cohort ((1) SDC, (2) ACC) evaluable for response. If 0 responses out of the first 9 evaluable patients are observed, the study will be stopped. In any other situation, the study will be continued until 17 patients are evaluable for response per cohort. If ≤2 responses are observed the study will accept the null hypothesis. If >2 responses are observed, the null hypothesis will be rejected. In the third cohort (other SGC) 9 patients will be included to evaluate the efficacy of cabozantinib in other subtypes of c-MET positive SGC. Because different subtypes are included in this cohort, these results are hypothesis forming but will not be used for statistical analysis. Therefore, this study cohort will be closed after the first stage with 9 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cabozantinib (Experimental): cabozantinib 60 mg tablets OD
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — cabozantinib tablets (Cabometyx®) once daily until progressive disease, intolerable toxicity, or investigator and/or patient decision to withdraw for a maximum duration of 2 years.
  Other Names: cabometyx

SUMMARY:
Phase 2 clinical trial on the efficacy of cabozantinib in locally advanced, recurrent and/or metastatic salivary gland cancer patients.

DETAILED DESCRIPTION:
Rationale: Salivary gland cancer (SGC) is a rare cancer with 24 histological subtypes. Treatment options for locally advanced and/or metastatic SGC are limited. The tyrosine kinase inhibitor cabozantinib suppresses tumor growth, angiogenesis, and metastasis, and has been approved for renal cell carcinoma and thyroid cancer. Cabozantinib may also be of value in advanced SGC because c-MET, one of the targets of cabozantinib, is frequently overexpressed in SGC.

Objectives: To assess the objective response rate (ORR), progression free survival (PFS), overall survival (OS), duration of response (DoR), toxicity, and quality of life (QoL) of patients with advanced SGC treated with cabozantinib in 3 cohorts: salivary duct carcinoma (SDC), adenoid cystic carcinoma (ACC), other SGC's.

Study design: Single arm, single center, phase II clinical trial in 3 cohorts: ACC, SDC and other SGC's.

Study population: Patient with c-MET positive, locally advanced, recurrent, and/or metastatic SGC.

Intervention: Cabozantinib tablets 60 mg once daily until progressive disease, intolerable toxicity, or investigator and/or patient decision to withdraw for a maximum duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

Disease specific

* locally advanced, recurrent, and/or metastatic SGC (excluding sarcomas and mesenchymal tumors)
* c-MET positive disease
* Measurable disease per RECIST version 1.1 Cohort-specific criteria
* SDC cohort: direct inclusion (no objective tumor growth prior to inclusion needed)
* ACC cohort: inclusion after objective growth in the last three months or complaints due to the disease
* Other SGC's: inclusion after objective growth in the last three months or complaints due to the disease General conditions
* Age ≥18 years
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Normal number of neutrophils and thrombocytes
* Liver function: ALT and AST < 2.5 x upper limit of normal (ULN), total bilirubin ≤ 1.5 x ULN (except for Gilbert's syndrome), serum albumin ≥28 g/L
* Renal function: creatinine < 1.5 x ULN or calculated creatinine clearance ≥ 40 ml/min, Urine protein/creatinine ratio ≤113.1 mg/mmol (≤1 mg/mg) or 24-hour urine protein <1 g
* Hemoglobin A1c (HbA1c) ≤ 8% or a fasting serum glucose ≤ 9 mmol/l

Exclusion Criteria:

General conditions

* A known allergy for cabozantinib or its components
* Long QT-syndrome
* Pregnancy or lactation
* Patients (M/F) with reproductive potential not implementing adequate contraceptives measures
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 3 months before inclusion
* Major surgery within 3 months before randomization. Complete wound healing from major surgery must have occurred 1 month before inclusion and from minor surgery at least 10 days before inclusion
* Uncontrolled illness including, but not limited to cardiovascular disorders including symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias, uncontrolled hypertension defined as sustained systolic BP > 150 mm Hg, or diastolic BP > 100 mm Hg, stroke (including TIA), myocardial infarction, or other ischemic event within 6 months before inclusion, serious active infections Concomitant treatments
* Concomitant (or within 4 weeks before inclusion) administration of any other experimental drug under investigation.
* Concurrent treatment with any other anti-cancer therapy.
* Concomitant anticoagulation. Low dose aspirin for cardioprotection and low dose LMWH are permitted.
* Radiation therapy within the last 4 weeks before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
overall response rate | every 8 weeks (first year of treatment) and every 12 weeks (second year of treatment) a CT/MRI scan will be made to asses the response rate until progressive disease
  Response will be measured according to RECIST version 1.1, the overall response rate is defined as the sum of the complete remissions plus partial responses. The best response will be used in each patient

SECONDARY OUTCOMES:
progression free survival | every 8 weeks (first year of treatment) and every 12 weeks (second year of treatment) a CT/MRI scan will be made to asses PFS until progressive disease
  progression free survival is defined as time from study enrollment until disease progression or death. Outcome will be scored as 'progressed' or 'censored' according to the FDA guidance for industry of clinical trial endpoints.
overall survival | Every OPD visit (starting with every 2 weeks, increasing to every 12 weeks after 1 year)
  overall survival is defined as time from study enrollment until date of death of any cause. Analysis of OS will be done at the end of the study (study related follow-up will be until 3 years after start of treatment)
duration of response | every 8 weeks (first year of treatment) and every 12 weeks (second year of treatment) a CT/MRI scan will be made to asses duration of response until progressive disease
  duration of response is defined as time from study enrollment until date of documented tumor progression or death. Only patients with a CR or PR will be included in the assessment of duration of response.
clinical benefit rate | every 8 weeks (first year of treatment) and every 12 weeks (second year of treatment) a CT/MRI scan will be made to asses the clinical benefit rate until progressive disease
  defined as the sum of complete remissions, partial responses, and patients with stable disease for >6 months.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion. At every visit AE's will be recorded. Scheduled visits will be planned 2, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 56, 68, 80, 92 and 104 weeks after start of treatment
  adverse events will be reported as descriptive statistics in a table
quality of life based on the EORTC QLQ-C30 questionnaire | patients are asked to fill in the questionnaires in week 0 (before start of treatment), week 8, 16, 24, 40, 56, and at progressive disease (up to 104 weeks after start of study medication).
quality of life based on the EORTC QLQ-H&N35 questionnaire | patients are asked to fill in the questionnaires in week 0 (before start of treatment), week 8, 16, 24, 40, 56, and at progressive disease (up to 104 weeks after start of study medication).
quality of life based on the PSSHN questionnaire | patients are asked to fill in the questionnaire in week 0 (before start of treatment), week 8, 16, 24, 40, 56, and at progressive disease (up to 104 weeks after start of study medication)..
pain level assessed by the VAS(visual analog scale) questionnaire | patients are asked to fill in the questionnaire in week 0 (before start of treatment), week 8, 16, 24, 40, 56, and at progressive disease (up to 104 weeks after start of study medication).
  scale range 0-10, in which a higher score represents more pain
response rate with continues tumor shrinkage end-points | every 8 weeks (first year of treatment) and every 12 weeks (second year of treatment) a CT/MRI scan will be made to asses the response rate until progressive disease
  response rate depicted in a waterfall plot
circulating tumor DNA levels | circulating tumor DNA levels will be measured at baseline, at week 2, week 4 and before every evaluation CT/MRI scan.
  circulating tumor DNA levels will be assessed to evaluate whether treatment response and disease progression can be predicted.
correlation of c-MET immunohistochemical score with treatment response | c-MET will be measured once (before treatment). Response will be measured every 8 weeks (first year) and every 12 weeks (second year of treatment)
  c-MET immunohistochemical score ranges from 0 to 300.

CONTACTS AND LOCATIONS:
Overall Officials: Carla ML van Herpen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weijers JAM, de Bitter TJJ, Verhaegh GW, van Boxtel W, Uijen MJM, van Engen-van Grunsven ACH, Driessen CML, Schalken JA, Ligtenberg MJL, van Herpen CML. Exploring the potential of circulating tumour DNA to monitor treatment response in salivary duct carcinoma patients of the CABO-ASAP trial. Oral Oncol. 2023 Dec;147:106620. doi: 10.1016/j.oraloncology.2023.106620. Epub 2023 Nov 6. No abstract available. PMID 37939426
- [Derived] van Boxtel W, Uijen MJM, Krens SD, Dijkema T, Willems SM, Jonker MA, Pegge SAH, van Engen-van Grunsven ACH, van Herpen CML. Excessive toxicity of cabozantinib in a phase II study in patients with recurrent and/or metastatic salivary gland cancer. Eur J Cancer. 2022 Jan;161:128-137. doi: 10.1016/j.ejca.2021.10.033. Epub 2021 Dec 14. PMID 34920917

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT03729297/Prot_SAP_000.pdf